CLINICAL TRIAL: NCT00615888
Title: Prospective Randomized Controlled Trial to Evaluate Fast Track Recovery in Elective Open Infrarenal Aortic Aneurysm Repair
Brief Title: Fast Track Management in Elective Open Infrarenal Aortic Aneurysm Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Bernd Muehling, M.D., Department of Thoracic and Vascular Surgery, University of Ulm, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119/2005
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2005-09

CONDITIONS: Aortic Aneurysm
Keywords: elective open repair; complications; morbidity and mortality; fast track patient management
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Traditional management including preoperative bowel washout, patient controlled analgesia (PCA), delayed start of enteral feeding
  Interventions: Procedure: Traditional management
- B (Experimental): Fast track management including no bowel washout, patient controlled epidural anesthesia, early enteral feeding
  Interventions: Procedure: Fast track patient management

INTERVENTIONS:
Procedure: Fast track patient management — no bowel washout, patient controlled epidural anesthesia, early enteral feeding
  Arms: B
Procedure: Traditional management — preoperative bowel washout, patient controlled analgesia, delayed start of enteral feeding
  Arms: A

SUMMARY:
Fast track programs have been introduced in many surgical fields to minimize postoperative morbidity and mortality. Morbidity after elective open infrarenal aneurysm repair is as high as 30%, mortality ranges up to 10%. In terms of open infrarenal aneurysm repair no randomized controlled trials exist to introduce and evaluate such patient care programs.

DETAILED DESCRIPTION:
Prospective randomization of patients admitted with infrarenal aortic aneurysm who undergo elective open repair in a "traditional" and "fast track" treatment arm. Main differences consist in preoperative bowel washout (none vs. 3L cleaning solution) and analgesia (patient controlled analgesia vs. patient controlled epidural analgesia: PCA vs. PCEA). Study endpoints are morbidity and mortality, need for postoperative mechanical ventilation and length of stay (LOS) on intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* infrarenal aortic aneurysm
* given written informed consent

Exclusion Criteria:

* contraindication for epidural anesthesia
* suprarenal clamping

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2007-10 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality after open infrarenal aortic aneurysm repair | 2 years

SECONDARY OUTCOMES:
LOS of ICU treatment, need for postoperative mechanical ventilation, day of discharge | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ulm, Ulm, Germany

REFERENCES:
- [Derived] Muehling BM, Ortlieb L, Oberhuber A, Orend KH. Fast track management reduces the systemic inflammatory response and organ failure following elective infrarenal aortic aneurysm repair. Interact Cardiovasc Thorac Surg. 2011 May;12(5):784-8. doi: 10.1510/icvts.2010.262337. Epub 2011 Feb 22. PMID 21343153
- [Derived] Muehling B, Schelzig H, Steffen P, Meierhenrich R, Sunder-Plassmann L, Orend KH. A prospective randomized trial comparing traditional and fast-track patient care in elective open infrarenal aneurysm repair. World J Surg. 2009 Mar;33(3):577-85. doi: 10.1007/s00268-008-9892-2. PMID 19137363